CLINICAL TRIAL: NCT05650125
Title: PINCER (A Platform Study for solId orgaN CancERs); an Agile Regional Platform Study to Deliver High Quality Translational Research
Brief Title: A Platform Study for solId orgaN CancERs
Acronym: PINCER
Status: Recruiting | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Countess of Chester NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Clatterbridge Centre for Oncology (Other); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Liverpool Womens Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 174008
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Surgery
Keywords: Surgery; Cancer; Translational; Biosample; Cohort
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary & metastatic tumour (biopsy/resection) - FFPE, fresh tissue, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with solid organ cancer: Prospective biosampling of blood/tissue
  Interventions: Other: Biosampling

INTERVENTIONS:
Other: Biosampling — Biosampling of blood/tumour/adjacent normal tissue

SUMMARY:
Generating bespoke biosampling protocols for individual tumour specific translational projects is onerous, cumbersome and inefficient. This study aims to provide a broad platform to maximise the unique access to biopsy and resected tumour specimens available from cancer patients to provide a high-quality and efficient source of biosamples for specific translational projects. Access to historical FFPE samples and clinical data, as well as prospective fresh tissue samples, will allow interrogation of the underlying biology of these cancers. Matched pseudoanonymised clinical and radiological data will allow the development of rich high-yield datasets.

DETAILED DESCRIPTION:
This is a platform tissue collection study to provide biosamples for specific research projects. These sub-studies will be proposed by interested researchers and undergo internal review by the PINCER steering committee. Following approval, each sub study will be delivered on this platform in line with this protocol. This study will not be used to generate biobanks, but to allow biosamples to be used for specific active sub studies.

1. Study Locations & Approval This platform will allow patients having surgery or biopsy for any solid organ cancer to consent to take part in the study. Any site wishing to do this will open as a site for the PINCER Study. Sub-studies using PINCER will require their own local study lead and SOP written by the local team and this will require approval by the PINCER steering committee. This will be to confirm alignment with the overarching PINCER protocol, define sampling requirements and assess the scientific validity of the study, as well as ensure regulatory oversight.
2. Fresh Tissue Collection Tissue will be obtained either through biopsy (an extra sample of tissue will be taken using the same needle at the time of original biopsy) or after surgical resection (where the tumour tissue would routinely be discarded after sampling for pathological assessment). In the case of tissue retrieved after surgery, a pathologist will ensure that excess tissue removed after resection will not compromise pathological assessment of the resected specimen.

   At the same time as biopsy or surgery, a small sample of blood (60ml) may be removed from the venous catheter which the patient has inserted as part of the routine care during their procedure. After the tissue has been retrieved, tissue and blood will be transported to a HTA approved facility. This will be performed under a locally arranged material transfer agreement (MTA) agreed by the local team between each individual site and the relevant partner organization.
3. Collection of historical FFPE tumour tissue Patients who have undergone biopsy or surgery for solid organ cancers will be identified from existing NHS clinical databases which track surgical activity by relevant clinical teams. Their tumour tissue samples will then be identified using local pathology systems, and their archived tissue blocks retrieved. In the case of patients who have had metastatic disease resected, both primary and metastatic tumour tissue will be accessed. A small amount of these tissue blocks will be sampled, and the remnant tissue block returned to the pathology archive. After the tissue has been retrieved, it will be transported to a HTA approved facility. This will be performed under a locally arranged material transfer agreement (MTA) between each individual site and the relevant partner organization.
4. Collection of post-treatment blood samples Up to 60mls of blood may be drawn from patients up to 12 months following treatment. After the blood has been retrieved, it will be transported to a HTA approved facility. This will be performed under a locally arranged material transfer agreement (MTA) between each individual site and the relevant partner organization.
5. Quality of Life Analysis Where appropriate, patients will be invited to complete EORTC Quality of Life assessment questionnaires up to 12 months following treatment.
6. Pseudoanonymised data & radiology collection Linked clinicopathological and radiological data will be retrieved where appropriate and stored on password protected computer systems. Local pseudoanonymisation will be required before these data are shared with other researchers not directly involved in the clinical care of patients.
7. Biosample analysis All analyses will be performed in HTA approved laboratories or equivalent. Pseudoanonymised samples may be shared with academic and commercial partner organisations within the UK and abroad, including the USA. All users of biosamples will be expected to have completed MRC HTA training.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy or surgical resection as standard of care

Exclusion Criteria:

* Refusal or inability to consent, paediatric patients

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a solid organ malignancy requiring surgery or biopsy as part of their routine clinical care as decided by the specialist MDT.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Biosample procurement | 4 years
  Patient biosamples delivered via platform

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pseudoanonymised linked clinical data will be available on request by translational researchers